CLINICAL TRIAL: NCT00312325
Title: Effect of High-Dose Prednisolone (Solu Dacortin®) Treatment on Choroidal and Optic Nerve Head Blood Flow in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPHT-030602
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2006-04-10 (Estimated); Status verified 2006-03

CONDITIONS: Regional Blood Flow; Optic Disk
Keywords: Optic nerve head blood flow; Choroidal blood flow; Prednisolone; Graves´ Ophthalmopathy; optic neuritis
MeSH Terms: conditions — Graves Ophthalmopathy; Optic Neuritis | interventions — Prednisolone

INTERVENTIONS:
Drug: Prednisolone

SUMMARY:
Because of their antiinflamatory effects, glucocorticoids are often used to reduce edema in neurologic tissue and to otherwise mitigate the consequences of neural inflammation. For example, high dose prednisolone treatment has been shown to be an effective therapy for different eye diseases including severe Graves´ Ophthalmopathy and acute optic neuritis. However, contradictory results exists for the influence of high dose prednisolone therapy per se on tissue blood flow. Thus, in the current study, we plan to investigate the effect of high dose, short time therapy with intravenous prednisolone in patients with optic neuritis and severe Graves´ Ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 and 65 years, nonsmokers
* Group A: Patients with Graves´ Ophthalmopathy (moderate to severe and active ophthalmopathy; i.e. clinical activity score >3 or =3) suitable for high-dose treatment with prednisolone as assessed by an independent ophthalmologist
* Group B: Patients with acute onset of optic neuritis suitable for high-dose treatment with prednisolone suitable for high-dose treatment with prednisolone as assessed by the ophthalmologist
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant and not to interfere with prednisolone treatment (normal liver blood parameter and hepatitis serology).
* Ametropy of less than 3 dpt.

Exclusion Criteria:

* Regular use of medication which could interfere with the study objectives, especially treatment with vasoactive drugs
* Active peptic ulcer or insulin dependent diabetes mellitus
* Hepatitis or elevated hepatic blood parameters
* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Non invasive measurement of optic nerve and choroidal blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria